CLINICAL TRIAL: NCT06786832
Title: Characterization, Treatment, and Long-term Follow-up of Fatigued Patients in Primary Care
Acronym: iFAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Academic Primary Health Care Centre, Region Stockholm (Unknown)
Responsible Party: Principal Investigator, Elin Lindsäter, clinical psychologist, PhD, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-05857-01; STY-2023/0008 (Other Grant/Funding Number: FORTE); 2023-05920 (Other Grant/Funding Number: VR); 20240093 (Other Grant/Funding Number: AFA)
Record Dates: First submitted 2025-01-13; First posted 2025-01-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Fatigue; Fatigue Post Viral; Exhaustion Disorder; Fatigue Symptom; Fatigue Related to Cancer Treatment
Keywords: Psychological treatment; Primary care; cognitive behavioral therapy; blended treatment; randomized controlled trial; Fatigue; burnout; chronic stress; register data; cognitive testing
MeSH Terms: conditions — Fatigue; Burnout, Psychological | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavioral therapy for persistent fatigue (Experimental): The treatment consists of three main phases: 1) goal-setting; stabilizing sleep-wake patterns and even distribution of activities over the day (pacing). Attention-shifting and cognitive reappraisal 2. Gradual increase in physical activity followed by gradual increase in mental and social activity 3. Gradual steps to reach individual goals.
  Interventions: Behavioral: Cognitive behavioral therapy for persistent fatigue
- Care as usual (CAU) (Other): Since there are no standardized, structured care programs and guidelines for the patient group, CAU may include a broad variety of psychosocial support, psychological treatment, physiotherapy, occupational therapy, pharmacological treatment, follow-up within specialist healthcare, and/or follow-up by general practitioners. An important aim of the project is to carefully map the content and scope of the care offered to patients in the study within the framework of CAU.
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for persistent fatigue — The treatment is based on a treatment manual that has previously been evaluated in several randomized controlled trials for persistently fatigued patients with various types of chronic somatic disorders (primarily in specialized healthcare settings).
  In this trial we have translated the treatment manual to Swedish and adopted it for implementation in a Swedish primary care setting. The treatment format is "blended", meaning that the treatment is administered both via an online platform (where the participant can communicate with the therapist through asynchronous text-messages) and via face-to-face therapy sessions with the therapist.
  Other Names: iFAS
  Arms: Cognitive behavioral therapy for persistent fatigue
Other: Care as usual — Since there are no standardized, structured care programs and guidelines for the patient group, CAU may include a broad variety of psychosocial support, psychological treatment, physiotherapy, occupational therapy, pharmacological treatment, follow-up within specialist healthcare, and/or follow-up by general practitioners. An important aim of the project is to carefully map the content and scope of the care offered to patients in the study within the framework of CAU.
  Other Names: CAU
  Arms: Care as usual (CAU)

SUMMARY:
The overarching purpose of this project is to further the understanding of fatigue as a symptom in primary care patients, and to build evidence for a highly accessible treatment targeting fatigue that can be readily implemented in primary care clinics.

Data will be collected within a randomized controlled superiority trial (RCT; N = 500). The primary aim is to evaluate the effectiveness of a novel cognitive behavioral therapy (iFAS: Internet-delivered treatment of Fatigue Across Syndromes) for fatigued patients as compared to care as usual (CAU). Primary outcome will be change in fatigue severity (as measured by the Checklist Individual Strengths, fatigue subscale) pre- to post-treatment (6 months), with long-term controlled follow-up after 12 months. A registry-based follow-up will be conducted up to 60 months post baseline. Moderators and mechanisms of treatment effect will be investigated with the aim to identify potential subgroups of fatigued individuals across and within diagnostic categories that may respond differently to treatment. Lastly, a health economic evaluation of long-term treatment effects will be conducted, which incorporates much needed detailed mapping of care as usual for fatigued patients.

DETAILED DESCRIPTION:
Background:

Fatigue can be defined as extreme and persistent tiredness, weakness, or exhaustion that that could be mental physical, or both. Fatigue is associated with increased healthcare consumption, work disability, and excess mortality, and has been studied extensively under different labels since the 1800's (e.g., neurasthenia, burnout, chronic fatigue syndrome). Studies in primary care populations indicate that about 20-30% of patients report fatigue, with up to 10% of patients presenting with fatigue as their main complaint. Although often considered a disorder-specific characteristic, the etiology and pathogenesis of fatigue are largely unknown and are generally believed to be multifactorial. No biological markers or other objectively measurable factors (such as cognitive impairment) have been found thus far that consistently and sufficiently explain the onset and perpetuation of disorder-specific fatigue. The high prevalence and non-specific nature of fatigue presents a challenge to general practitioners who generally have limited time and resources for assessment and intervention.

Importantly, a potential break-through to how we can understand fatigue has been achieved in recent years, with studies showing that variance in fatigue severity is better explained by transdiagnostic factors (i.e., factors not attributable to a specific medical condition, such as demographic and psychosocial variables and aspects of daily functioning) than by disorder-specific pathophysiology. Further, similar cognitive and behavioral perpetuating mechanisms of fatigue (such as fear avoidance, symptom catastrophizing, self-efficacy, and resting-behavior) have been found across disorders. These findings suggest that a transdiagnostic approach to understanding and treating persistent fatigue might be beneficial for patients and healthcare practitioners, with potentially important implications for treatment.

Treatment of fatigue:

As with other aspects of fatigue, intervention research on fatigue has primarily been conducted in disorder-specific pipelines using disorder-specific protocols. CBT is the most studied treatment, with promising effects for patients with, for example, chronic fatigue syndrome, post-infectious fatigue, and various long-term medical conditions where fatigue is often central (both face-to-face and when delivered via the internet; ICBT). Results from previous RCTs conducted by the investigators have indicated that CBT can be an effective treatment to reduce symptom burden in patients diagnosed with stress-induced exhaustion disorder. Importantly, disorder-specific CBT-protocols for fatigue are largely similar across clinical groups, and the same cognitive and behavioral responses to fatigue have been found to moderate and mediate fatigue severity after CBT across a range of fatigued patient groups.

Even though CBT may hold promise to reduce fatigue severity in different clinical groups, many fatigued patients still do not receive treatment, and not all patients who receive CBT are sufficiently helped. Further research is needed to understand symptom presentation and development as well as treatment moderators, predictors, and mediators of change. Also, there is a significant knowledge gap regarding how fatigue can be identified and treated in an early phase in the primary care context. Given the similarities in effective treatment protocols across fatigued samples, together with potentially common change mechanisms, investigating the effectiveness of a transdiagnostic treatment protocol is a promising avenue with enormous potential utility to increase clinical effects, accessibility, and large-scale implementation. To date, no transdiagnostic treatment specifically targeting fatigue across patient groups has been evaluated.

The current study:

Based on previous disorder-specific treatment protocols aimed to reduce fatigue severity in various fatigued populations, the investigators have developed a transdiagnostic intervention adapted for primary care patients who suffer from persistent fatigue independent of primary diagnosis (iFAS: Internet-delivered treatment of Fatigue Across Syndromes). The treatment is delivered in a blended format (face-to-face therapy combined with internet-delivered texts and exercises) and is administrated over 4 - 6 months. The feasibility of iFAS has recently been evaluated in a non-randomized feasibility trial (Clinical trials ID: NCT06341751).

Study design:

The planned study is a randomized clinical superiority trial that will recruit fatigued patients listed at primary healthcare clinics in Region Stockholm. Study participants (N=500) will be randomized to iFAS (n=250) or to CAU (n=250) by a person not related to the study. Due to the nature of the study, blinding to treatment condition will not be possible.

Data collection includes clinician-rated data, self-rated symptom measures, and registry data using interlinked microdata from regional and national registers. Cognitive functioning will be assessed using a digital cognitive test-battery that will be administered at baseline and at the 12-month follow up. Additionally, the study will explore changes in physiological variables (in a subset of participants) from baseline to the 12-month follow-up using continuous data collected from biometric rings.

Research questions:

RQ1. Is iFAS associated with a greater post-treatment reduction in fatigue severity (primary outcome) and secondary outcome domains (self-rated symptoms, cognitive functioning, net days on sick leave) compared to CAU?

RQ2. What characterizes the fatigued sample at baseline in terms of sociodemographic, clinical, and biometric variables? Can clinically relevant subgroups of patients be identified that share similar characteristics?

RQ3. Which factors moderate and mediate the effect of iFAS vs. CAU and which factors predict symptom development? We hypothesize (1) that there will be transdiagnostic subgroups of patients that differ in treatment response based on baseline characteristics as identified in RQ2, that (2) these characteristics can be used to model treatment outcomes using supervised machine learning, and further that (3) changes in cognitive and behavioral responses to fatigue (e.g., fear avoidance, catastrophizing about symptoms, all-or-nothing behavior) as well as sleep- and physical activity patterns will mediate the effect of iFAS vs. CAU.

RQ4. Are there differences between participants who received iFAS vs. CAU at the 12- and 60-month follow-up and do individual characteristics moderate these differences?

RQ5. Is iFAS vs. CAU a cost-effective treatment at the 12 month follow-up? Indirect (e.g., work absenteeism, sick leave) and direct (e.g., healthcare consumption) costs will be evaluated using data from national registers.

RQ6. Which healthcare interventions are provided for participants who are randomized to CAU, and do sociodemographic, geographic, and clinical factors predict the type and extent of treatment delivered?

Recruitment procedure:

This study will recruit participants directly from primary care clinics in Region Stockholm. Hence, no advertisement in newspapers or in social media will be conducted to target potential study participants. All information about the study, aimed at both study participants and primary care staff, will be made available on a study webpage.

Patients can be referred to the study by their primary care physician if they (a) report at least three months of persistent, functionally disabling fatigue as a central symptom and (b) the general practitioner (GP) has assessed that the fatigue is not a direct effect of an active disease process motivating another treatment (e.g., hypo-/hyperthyroidism, anemia, cancer, dementia, sleep apnea, post-traumatic stress disorder) or a side-effect of medication. See below ("Eligibility") for inklusion/exclusion criteria.

Estimated sample size and power:

For 90% power to detect a standardized between-group effect size of d=0.25 on the primary outcome (α=.05), an intraclass correlation between measurements of 0.7, and an expected attrition of 20%, 250 patients will be included in each arm (total sample size: N=500).

Statistical methods:

Analyses will be based on an intention-to-treat approach. Change in the primary outcome measure will be analyzed using mixed effects linear regression. Change from baseline to treatment completion (6 months post baseline) will be the primary endpoint. Fixed predictors in these analyses will be time, group and their interaction effect while taking individual variation in baseline symptom levels and change over time into account (i.e., random intercept and/or slope).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-67
2. enrollment at a primary care clinic in Region Stockholm
3. severe, functionally disabling fatigue as a central symptom for at least 3 months
4. The fatigue has an identifiable start and hence has not been life-long;
5. The fatigue is not a direct effect of an active disease process motivating another treatment (e.g., hypo-/hyperthyroidism, anemia, cancer, dementia) or the effect of medication
6. regular access to a computer and to the Internet
7. ability to read and write in Swedish.
8. ability to visit a study center for participation in potential assessments and treatment sessions (maximum 60 minutes) and to take part of written material via the internet.

Exclusion Criteria:

1. substance abuse disorder in the past 6 months
2. Current or past psychosis or bipolar disorder
3. Primary psychiatric disorder of such severity that it merits evidence-based treatment (e.g., obsessive compulsive disorder, moderate to severe depression, post-traumatic stress disorder, anorexia nervosa)
4. elevated risk for suicide
5. deliberate self harm in the past 6-months (e.g., cutting, burning, poisoning);
6. BMI>40
7. Initiated or changed psychopharmacological medication (e.g., for depression or anxiety disorders) in the past month
8. ongoing chemotherapy
9. intellectual disability (e.g., severe autism) that affects ability to work with the treatment
10. pregnancy
11. life circumstances that complicate or make treatment impossible (e.g., domestic violence, ongoing legal disputes, disputes with social insurance agency, planed or on-going work capacity assesment regarding permanent work disability pension or planed surgery)
12. ongoing psychological treatment and/or multimodal rehabilitation.
13. working night shifts

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Self-rated fatigue severity | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline))
  Fatigue severity (self-rated) using the Checklist Individual Strengths - Fatigue severity subscale (CIS-F). The domain Fatigue severity contains 8 items scored on a 7-point Likert scale (range 8-56; higher scores=more severe fatigue).

SECONDARY OUTCOMES:
Concentration | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline)
  Concentration is a subscale in the Checklist Individual Strengths (CIS). The subscale contains 5 items scored on a 7-point Likert scale. Higher ratings indicate more problems with concentration.
Motivation | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline)
  Motivation is a subscale in the Checklist Individual Strengths (CIS). The subscale contains 4 items scored on a 7-point Likert scale. Higher ratings indicate more difficulties with motivation.
Activity | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline)
  Activity is a subscale in the Checklist Individual Strengths (CIS). The subscale contains 3 items scored on a 7-point Likert scale. Higher ratings indicate reduced activity.
Self-rated depressive symptoms | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months). Suicide-item will be administered every three weeks during the treatment phase.
  Patient Health Questionnaire-9 (PHQ-9). Scale range is from 0 to 27, higher scores representing more depressive symptoms. NOTE: The suicide-item will be administered every three weeks during the treatment phase).
Somatic symptoms | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  Physical Health Questionnaire-15 (PHQ-15). Scale range is from 0 to 30, higher scores representing more somatic symptoms
General anxiety | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  The General Anxiety Questionnaire (GAD-7). Scale range is from 0 to 21, higher scores representing more anxiety.
Insomnia Severity | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline)
  The Insomnia Severity Inventory (ISI) 7 items. Scale range is from 0 to 28, higher scores representing higher insomnia severity.
  An additional item will be added to assess hypersomnia.
Perceived Stress | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  The Perceived Stress Scale (PSS-10). Scale range is from 0 to 40, higher scores representing a higher level of perceived stress.
Burnout | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  The Shirom-Melamed Burnout Questionnaire (SMBQ-18). Scale range is from 0 to 6, higher scores representing a higher level of burnout.
Self-rated health | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  The Self-rated health questionnaire (SRH-5). A single item with 5 response-categories, 0 (very bad health); 4 (very good health)
Cognitive and behavioral responses to symptoms | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline)
  Process measure: Cognitive and behavioral responses to symptoms questionnaire (CBRQ), 18-items. The scale assesses six domains: Fear avoidance (3 items, scale range 0-12); Damage beliefs (3 items, scale range 0-12); Embarrassment avoidance (3 items, scale range 0-12); Symptom focusing (3 items, scale range 0-12); All-or-nothing behaviour (3 items, scale range 0-12); Resting behaviour (3 items, scale range 0-12).
General self-efficacy | Baseline (Pre intervention), during treatment phase (every three weeks), post (6 months after baseline) and long term follow up (12 months after baseline)
  Process measure: The General self-efficacy scale (GSE), 10 items. Scale range is from 10 to 40, higher scores representing a higher level of self-efficacy.
Functional disability | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), 12 items. Scoring from 0 (maximum functional disability) to 100 (no functional disability)
Work and Social Adjustment | Baseline (Pre treatment), Post treatment (6 months), long-term follow-up (12 months).
  The Work and Social Adjustment Scale (WSAS), 5 items. Scale range 0 to 40 with higher scores representing better work and social adjustment.
Self-rated exhaustion disorder (s-UMS) | Baseline, post treatment (6 months) and 12-month follow-up from baseline.
  s-UMS is a questionnaire developed for self-assessment of diagnostic criteria for exhaustion disorder. Eight diagnostic items are responded to as "yes" or "no". The last item pertains to consequences and functional disability and is responded to on a scale of 0 (no functional disability), 1 (yes, some functional disability), or 2 (yes, significant functional disability).
Symptoms of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) | Baseline, post treatment (6 months) and 12-month follow-up from baseline.
  A 25-item self-rated symptom questionnaire in which respondents first respond yes/no to each symptom and then in a second step, if "Yes", respond to the severity level of that symptom on a scale from 1-4 ("mild", "moderate", "severe", "very severe").
  Scores of symptom severity are added for a scale range of 1-100 (higher scores indicate higher symptom severity).

OTHER OUTCOMES:
Treatment credibility | Three weeks after treatment start
  Assessed using the Credibility/Expectancy Questionnaire (C-Scale). The C-Scale is a 5-item measure, scale range is 0 to 50 points with higher scores indicating higher treatment credibility.
Patient satisfaction with treatment/healthcare | Post-treatment (6 months)
  Client Satisfaction Questionnaire (CSQ-8). Total scores range from 8 to 32, with higher scores indicating greater treatment satisfaction.
  A slightly revised version will be administered to participants in the CAU group to probe satisfaction with healthcare.
Working alliance | Week 3 and 15 of treatment
  Assessed using the Working Alliance Questionnaire (WAI - short version). Scale range is from 6 to 42 with higher scores indicating a better percieved working alliance. Will only be administered to the exerimental treatment arm (iFAS)
Negative effects of treatment | Post treatment (6 months from baseline)
  The Negative Effects of Treatment Questionnaire (NEQ-20). The self-report measure consists of three parts. First, respondents endorse specific items in case they have occurred or not during treatment, yes/no (dummy coded as a variable: 1/0). Second, the respondents rate how negatively the negative effect was on four-point Likert-scale, ranging from "Not at all" to "Extremely", 0-4 ("0" being minimum and "4" being maximum). Third, the respondents attribute the negative effect to "The treatment I received" (1) or "Other circumstances" (0) (dummy coded as a variable: 1/0).
  A slightly revised version will be administered to participants in the CAU group to probe negative effects of healthcare.
Adverse events related to study participation/treatment | weeks 6, 12, 18
  Open-ended questions regarding potential adverse events will be administered to study participants in both treatment arm every 6 weeks during the treatment phase.
Cognitive functioning | Baseline and 12-month follow-up from baseline
  Will be assessed using a validated digital cognitive test battery. The test will assess attention and processing speed, executive functioning, and memory. The total test takes approximately 25 minutes to complete.
Healthcare consumption | Data will be collected from two years before inclusion in the study up to 60 months after inclusion, meaning from 2023-2030.
  Data will be collected from Region Stockholm's database (VAL) that provides information about all publicly funded outpatient and inpatient healthcare provided in Stockholm County, including number of healthcare visits.
Sickness absence | Data will be collected from two years before inclusion in the study up to 60 months after inclusion, meaning from 2023-2030.
  Data on sickness benefits as well as sickness and activity compensation will be retrieved from the Swedish Social Insurance Agency's database (MiDAS).
Individual-level socioeconomic information | Data will be collected from two years before inclusion in the study up to 60 months after inclusion, meaning from 2023-2030.
  Data will be retrieved from Statistics Sweden's LISA database (Longitudinal Integration Database for Health Insurance and Labour Market Studies) and include information about occupation and type of income and benefits.
Medication use | Data will be collected from two years before inclusion in the study up to 60 months after inclusion, meaning from 2023-2030.
  Registry data: National Board of Health and Welfares registry
  From the Prescribed Drug Register: Dispensed prescribed medications (ATC codes, dates, DDD).
Cause of death | Data will be collected from two years before inclusion in the study up to 60 months after inclusion, meaning from 2023-2030.
  Registry data: National Board of Health and Welfares registry
  From the Cause of Death register: (1) date of death and (2) causes of mortality.
Heart rate variability | Continuous data-collection from baseline to 12-month follow-up.
  A subset of participants will receive a non-invasive biometric ring (worn on participant finger) to collect data on heart rate variability from baseline to the 12-month follow up.
Sleep- and activity patterns | Continuous data-collection from baseline to 12-month follow-up.
  A subset of participants will receive a non-invasive biometric ring (worn on participant finger) to collect data on movement and sleep from baseline to the 12-month follow up.
Body temperature fluctuations | Continuous data-collection from baseline to 12-month follow-up.
  A subset of participants will receive a non-invasive biometric ring (worn on participant finger) to collect data on fluctuations in body temperature from baseline to the 12-month follow up.
Alcohol Use | Pre inclusion screening only
  AUDIT (Alcohol Use Disorders Identification Test) is used for screening for unhealthy alcohol use, defined as risky or hazardous consumption or any alcohol use disorder. It identifies alcohol intake, potential dependence on alcohol and, experience of alcohol-related harm.
Symptoms of autism | Pre inclusion screening only.
  The Ritvo Autism and Asperger Diagnostic Scale-Revised (RAADS-14) is a diagnostic tool specifically designed to assist in the identification of autism spectrum disorder (ASD) in adults. The scale ranges from 0-42 and covers three areas: Mentalizing deficits, Social anxiety and Sensory reactivity.
Symptoms of adhd in childhood | Pre inclusion screening only
  The Wender Utah Rating Scale - 25 item version (WURS-25) is a self-report instrument that is designed to retrospectively evaluate the presence and severity of childhood symptoms of ADHD in adults in the following areas: Impulsivity and Behavioural problems, Inattentiveness and School problems, Self Esteem and Negative mood. Scale ranges from 0-100 with scores above 36 indicating high likelihood of ahdh.
Hypermobility | Pre inclusion screening only
  The self-assessment five-part questionnaire on hypermobility (5PQ) consists of five items rated "Yes" or "No", with two or more "Yes" answers indicating generalised joint hypermobility.
Comorbidity (self-registered) | Pre inclusion screening only
  A list of 34 common somatic and psychiatric diagnosis known as the "Comorbidity table" was used. For each specific diagnosis the answers given are "No, never", "Yes, previous", and "Yes, ongoing".

CONTACTS AND LOCATIONS:
Overall Officials: Elin Lindsäter, PhD, Ass. Prof, Principal Investigator — Region Stockholm and Karolinska Institutet
Locations (1):
- Gustavsberg University Primary Care Clinic, Stockholm, Gustavsberg, Sweden

IPD SHARING:
Plan to Share IPD: No